CLINICAL TRIAL: NCT06293495
Title: Comparison of the Incidence of Cut-out Between Intramedullary Nails With Double Cephalic Screw vs. Unique in Pertrochanteric Fractures: a Prospective Randomized Clinical Trial
Brief Title: Incidence of Cut-out Using Intramedullary Nails With Double Cephalic Screw vs. Unique in Pertrochanteric Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Pedro-José Torrijos-Garrido, Principal Investigator, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUT-OUT
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Proximal Femoral Fractures
Keywords: Proximal femoral fracture; Hip fracture; Cut-out
MeSH Terms: conditions — Proximal Femoral Fractures; Hip Fractures

STUDY DESIGN:
Intervention Model Description: Randomized, prospective trial with a CE-marked medical devices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Cephalic Screw System (Active Comparator): A Gamma 3 nail (single cephalic screw system) will be used for osteosynthesis of the fracture.
  Interventions: Device: Gamma 3 Nail (Stryker)
- Double Cephalic Screw System (Experimental): A Chimaera nail (system with double cephalic screw) will be used for osteosynthesis of the fracture.
  Interventions: Device: Chimaera Nail (Orthofix)

INTERVENTIONS:
Device: Gamma 3 Nail (Stryker) — Open reduction an internal fixation of proximal femoral fracture with a Gamma 3 nail (single cephalic screw system)
  Arms: Single Cephalic Screw System
Device: Chimaera Nail (Orthofix) — Open reduction an internal fixation of proximal femoral fracture with a Chimaera nail (system with double cephalic screw)
  Arms: Double Cephalic Screw System

SUMMARY:
The goal of this clinical trial is to compare outcomes in the treatment of proximal femur fractures. The main question it aims to answer is whether the use of a double cephalic screw prevents nail failure (cut-out).

Participants will be treated using open reduction and internal fixation with a proximal femoral nail. Researchers will compare intramedullary nailing with a single cephalic screw (Gamma nail) and with a double cephalic screw (Chimaera nail) to see the cut-out rate.

DETAILED DESCRIPTION:
Randomized, open and prospective clinical trial.

Following the surgical indication for open reduction and internal fixation as treatment for proximal femoral fractures, patients will be randomly assigned (ratio 1:1) to one of the following treatments:

Control group: a Gamma 3 nail (single cephalic screw system) will be used for osteosynthesis of the fracture.

Experimental group: a Chimaera nail (system with double cephalic screw) will be used for osteosynthesis of the fracture.

Patient (or their legal guardian) must provide/sign the informed consent prior to inclusion in the study.

After the surgery, patients will be followed-up at 6 weeks, 3 and 6 months. At those times, data related to the radiological examination, the appearance of complications and the walking ability evaluation scale (FAC) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proximal femur fracture (OTA/AO 31-A1, A2 and A3) requiring surgical treatment.
* Signing of written informed consent according to current legislation before collecting any information, either by the patient or by the legal representative or by people linked by family ties.

Exclusion Criteria:

* Presence of other fractures in the ipsilateral femur that condition the surgical treatment of the pertrochanteric femur fracture.
* Subcapital fracture of the proximal femur.
* Subtrochanteric fracture of the proximal femur.
* Pathological fracture.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of cut-out. | 0-6 months
  Cut-out is a mechanical complication consisting of varus collapse and migration of the cephalic screw through the femoral head.

SECONDARY OUTCOMES:
Functional Ambulatory Categories (FAC) | 0-6 months
  Classifies patients into 6 categories based on their ability and need for assistance with ambulation. Classifies patients into 6 categories based on their ability and need for help with ambulation, where 0 is equivalent to a patient with the impossibility of ambulation and 5 is a patient completely independent for ambulation.
Tip-apex distance | 3-6 months
  Distance from the tip of the screw to the apex of the femoral head in the anteroposterior and axial views.
Parker index | 3-6 months
  Indicates the distance of the screw from the inferior edge of the femoral neck in anteroposterior view or from the posterior edge of the femoral neck in lateral view.
Baumgaertner reduction quality criteria | 3-6 months
  3 groups are established according to the quality of reduction: good, acceptable and bad
Number of Surgical complications (Intraoperative) | 0-1 month
  Intraoperative complications
Number of Surgical complications (post-operative) | 0-6 months
  Postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Pedro José Torrijos Garrido, MD, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No